CLINICAL TRIAL: NCT03205527
Title: Perturbation Training for Enhancing Stability and Limb Support Control for Fall-risk Reduction Among Stroke Survivors
Brief Title: Perturbation Training for Fall-risk Reduction Among Stroke Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Tanvi Bhatt, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0933; 1R01HD088543-01A1 (NIH)
Record Dates: First submitted 2017-06-23; First posted 2017-07-02 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Fall risk; Stroke survivors; Perturbation training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Slip training for chronic stroke (Experimental): Chronic stroke subjects in this training group will receive bilateral overground, slip perturbation training.
  Interventions: Other: Overground slip perturbation training
- Control for chronic stroke (No Intervention): Chronic stroke subjects, after baseline walking trials, will walk for about 30 trials at their preferred walking pace to match the total trials the other groups receive before receiving a single slip each randomly on their non-paretic and paretic sides.
- Slip training for sub-acute stroke (Experimental): Sub-acute stroke survivors in this training group will receive bilateral overground, slip perturbation training.
  Interventions: Other: Overground slip perturbation training
- Control for sub-acute stroke (No Intervention): Sub-acute stroke subjects, after baseline walking trials, will walk for about 30 trials at their preferred walking pace to match the total trials the other groups receive before receiving a single slip each randomly on their non-paretic and paretic sides.

INTERVENTIONS:
Other: Overground slip perturbation training — Slips will be induced by a low-friction platform (65×30×0.6 cm, μ<0.05) embedded side-by-side in the walking path, set nearly flush with the floor surround. The moveable platform, mounted on top of a pair of force platforms (AMTI, Newton, MA) for measuring ground reaction forces is firmly locked in a stationary position. An unannounced release occurs at heel strike of the perturbed, without the knowledge of subject, after which the platform is free to slide up to 150 cm. The mechanical release is controlled by the loading on the force platforms and the computer.
  Arms: Slip training for chronic stroke; Slip training for sub-acute stroke

SUMMARY:
The long-term objective of this research is to develop an efficacious training paradigm to enhance stroke survivors' defense mechanisms against falls and possibly reduce healthcare cost. The Centers for Disease Control and Prevention estimates the direct medical cost for fall related injuries to be $34 billion annually. Forty percent to 70% of community-dwelling stroke survivors experience detrimental falls each year and tend to have 1.5 to 4 times higher risk of hip fracture than their healthy counterparts; with only less than 40% of those individuals regaining independent mobility. Falls, thus not only affect activities of daily living but also reduce mobility, increase risk of second stroke and mortality. Despite potential financial and functional implications of falls in this population, health-care personnel are limited in their ability to develop and validate interventions to reduce fall-risk for them. Further emphasis is placed on locomotor training with focus on enhancing paretic limb function. The project design consists of a randomized controlled trial to examine the ability of chronic stroke survivors to acquire, generalize and retain adaptations to slip-perturbation training for not only mitigating fall risk but also improving walking function. It also explores translation of this paradigm to the sub-acute population. The paradigm is novel in that it targets contributions of the paretic vs. non-paretic limbs on fall-risk through a bilateral training paradigm that involves training the non-paretic side first and then paretic to facilitate acquisition of fall-prevention skills on the paretic side, which may otherwise take longer to acquire training effects. The longer-term benefits of such perturbation training, targeting both limbs for reducing falls will be assessed not only in the laboratory but also in real life via wearable sensors, along with improved community walking function. The hypothesis of this study if supported by the results will provide an evidence-supported training protocol to reduce the fall-risk not only in people living with hemiparetic stroke but also among survivors of other acquired unilateral cortical lesions.

DETAILED DESCRIPTION:
Approximately 800,000 Americans suffer a stroke every year and 689,450 reported having short and long-term disabilities leading to dependence in activities of daily living. It has been reported that stroke survivors experienced detrimental falls each year and most occurring during walking. The likelihood of experiencing a fall upon discharge from rehabilitation being significantly higher than during the rehabilitative phase. Falls resulting from environmental perturbations such as slips contribute to a significant percentage of these falls. Hence, it is important to develop innovative and effective paradigms for fall-risk reduction in chronic as well as sub-acute stroke survivors. The purpose of this research is to understand the effect of bilateral slip-perturbation training protocol targeting training both paretic vs. non-paretic limbs on fall-risk reduction and prevention. Also, to find its effect on increasing community ambulation in community dwelling stroke survivors.

Participants in this study will be individuals with chronic (> 6 months) hemiparesis following stroke or individuals with sub-acute stroke (> 6weeks and < 6 months), ambulatory (with or without assistive device) and more than 21 years of age. Subjects will be screened for the inclusion criteria. If subjects pass the screening, they will go through the full clinical balance assessment and laboratory dynamic stability test. The chronic stroke survivors will be randomized into two groups: - Group A: Slip training group; Group B: Control group. While, the sub-acute stroke survivors will be randomized into two groups: - Group C: Slip training group; Group D: Control group.

For the slip training groups (A and C), all subjects' normal walking pattern and their recovery responses to slip will be recorded with a motion tracking system (including videotaping) while they walk across an instrumented area along a straight path in the lab. A slip will be induced after a subject steps on a low-friction platform.

For the chronic stroke subjects, baseline activity monitoring using wearable sensors will be performed for up to four weeks prior to the training session followed by activity monitoring for 12 months. While for the sub-acute stroke subjects, it would be done for 6 months.

For groups A and B, the follow-up stability test will be at 6 and 12 months post-training session, which will consist only of one slip induced on the training side and contralateral side. For groups C and D, follow-up session is 6 months post training session.

Incidence of falls and physical activity will be monitored between training and re-test sessions through falls, activity monitoring-questionnaire to describe details of the falls and through the wearable sensors for groups A, B, C and D.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have to be ambulatory (with or without assistive device) with self-reported chronic (> 6 months) stroke-induced hemiparesis confirmed by participants' physician and medically cleared. Evidence of unilateral brain lesion confirmed by an imaging study (e.g. CT or MRI).
* Subjects with no other acute and significant neurological, cardiopulmonary, musculoskeletal or systemic diagnosis or have undergone a recent major surgery (<6 months) or hospitalization (<3 months) and not on any sedative drugs
* Ability to walk at least 10m with or without assistive device which includes use of ankle orthosis or functional electrical stimulation devices (which is equivalent to having a score of> 4, dependent supervision on Functional Ambulatory category scale)

Exclusion Criteria:

* Severe osteoporosis (Ultrasound score < -2)
* Cognitive impairment (Mini Mental State Exam score<25)
* Aphasia (<71% on Mississippi Aphasia Screening Test)
* Severe depression ( > 15 on Geriatric Depression Scale)
* Severe obesity (BMI >35Kilogram/m2)
* Complains of shortness of breath, or uncontrolled pain (> 3/10 on VAS), or if pulse oxygen drops <92% on the 6 minute walk test (for endurance)
* Uncontrolled hypertension (resting systolic blood pressure > 165 mmHg and/or diastolic blood pressure > 110mmHg)
* Resting heart rate > 85% of age-predicted maximal heart rate
* Resting oxygen saturation <95%

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in laboratory induced falls | Pre-training, immediate post-training, 6-month post training, 12-month post training
  Perturbation is induced successfully and safely to reproduce inadvertent falls in a protective laboratory environment. Falls will be measured by amount of force recorded on the load cell attached to the ceiling mounted safety harness system donned by the participant. Instability of the body's COM and poor limb support prior to touchdown of the recovery step account for 90~100% of subsequent falls (occurring ~500ms later) in both sit-to-stand-slip and in gait-slip, in the laboratory settings.
Change in real life falls | Retrospectively assessed via participant history for 12 months before pretest and prospectively assessed for 12 months post training via falls diary
  Real life falls are measured to determine if training effect can be translated into everyday real life setting.

SECONDARY OUTCOMES:
Change in Stability | Pre-training, immediate post-training, 6-month post training, 12-month post training
  Stability is defined by both the position of a person's center-of-mass (COM) with respect to his or her base-of-support (BOS) and it's velocity.
Change in Limb support | Pre-training, immediate post-training, 6-month post training, 12-month post training
  The inability to provide timely limb support due to insufficient amount of upward impulse generated from the ground reactive force can cause limb collapse, as characterized by the quotient of amount and rate of hip descent (Vhip/Zhip) measured from hip height and lead to an eventual fall.
Change in gait speed | Pre-training, 6-month post training, 12-month post training
  Gait speed will be computed from an average of three walking trials on the laboratory walkway.
Change in symmetry | Pre-training, 6-month post training, 12-month post training
  Symmetry will be computed from an average of three walking trials on the laboratory walkway.
Change in gait speed during functional ambulation | One month before pretest till prospectively 12 months post training
  The gait speed for each day will be calculated by patient's wearable sensor and their assistive device sensor. This parameter will be used to analyze improvement in ambulatory skills of the patient and decrease reliance on the assistive device.
Change in physical activity | One month before pretest till prospectively 12 months post training
  The total number of steps and distance for each day will be calculated by patient's wearable sensor and their assistive device sensor. This parameter will be used to analyze improvement in physical activity of the patient and decrease reliance on the assistive device.

CONTACTS AND LOCATIONS:
Overall Officials: Tanvi Bhatt, PhD PT, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhatt T, Dusane S, Gangwani R, Wang S, Kannan L. Motor adaptation and immediate retention to overground gait-slip perturbation training in people with chronic stroke: an experimental trial with a comparison group. Front Sports Act Living. 2023 Sep 13;5:1195773. doi: 10.3389/fspor.2023.1195773. eCollection 2023. PMID 37780126
- [Derived] Dusane S, Bhatt T. Can prior exposure to repeated non-paretic slips improve reactive responses on novel paretic slips among people with chronic stroke? Exp Brain Res. 2022 Apr;240(4):1069-1080. doi: 10.1007/s00221-021-06300-8. Epub 2022 Feb 1. PMID 35106605
- [Derived] Gangwani R, Dusane S, Wang S, Kannan L, Wang E, Fung J, Bhatt T. Slip-Fall Predictors in Community-Dwelling, Ambulatory Stroke Survivors: A Cross-sectional Study. J Neurol Phys Ther. 2020 Oct;44(4):248-255. doi: 10.1097/NPT.0000000000000331. PMID 32815890